CLINICAL TRIAL: NCT02749175
Title: Novel Ultrathin Miniature Force Sensor to Deliver Optimal Cricoid Pressure for Airway Protection in Patients at High Risk of Gastric Aspiration - a Verification of Design
Brief Title: SMART Study (Sellick's Maneuver Assisted Real Time) to Deliver Target Cricoid Pressure in Simulated Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Hee Hwan Ing, Senior consultant, KK Women's and Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KKWCH
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Aspiration of Gastric Contents
Keywords: cricoid pressure
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cricoid force sensor monitor system (Experimental): Nurse applied cricoid pressure with a sensor guided by monitoring Nurses instructed to apply cricoid pressure at target force of 20-30 Newtons.
  Interventions: Device: Cricoid force sensor monitor system
- Sham cricoid force sensor monitor system (Sham Comparator): Nurse applied pressure on a sham sensor with no monitor input. Nurses instructed to apply cricoid pressure at target force of 20-30 Newtons
  Interventions: Device: Sham Cricoid force sensor monitor system
- Current standard (No Intervention): Nurse applied cricoid force according to memory. Nurses instructed to apply cricoid pressure at target force of 20-30 Newtons

INTERVENTIONS:
Device: Cricoid force sensor monitor system — Comprise of a sensor and a monitor system
  Arms: Cricoid force sensor monitor system
Device: Sham Cricoid force sensor monitor system — Comprise of a sensor and a sham monitor system
  Arms: Sham cricoid force sensor monitor system

SUMMARY:
Cricoid force is applied during airway management to prevent pulmonary aspiration of regurgitated gastric contents. This force is usually applied by a nurse or anaesthesia assistant. Currently this is performed WITHOUT monitoring and the force applied is determined by the individual's "educated hand" that is derived from his/her experience from past training and practice. Studies have shown that the actual force applied by nurse and anaesthesia assistant is inconsistent and deviates from the optimal force. Under application of cricoid force results in ineffective cricoid pressure and the risk of pulmonary aspiration. Consequences of pulmonary aspiration include lung injury and infection, hypoxia, long Intensive Care Unit stay and even death. Over exertion of cricoid force results in distortion of the larynx (leading to difficult bag mask, difficult tracheal tube insertion and hypoxia). Preliminary results from previous study (IRB 2014/437/D), an observation crossover pilot was carried out comparing the amount of cricoid force applied by 16 nurses on manikin with and without direct feedback. Nurses were instructed to apply a range of force of 30-44 Newtons on a marked site on the neck region of manikin. A flexiforce load sensor was used. Unblinded nurses performed significantly better with feedback using the load sensor then blinded nurses. With Funding from a National grant, a real-time measurement of cricoid force is developed to give feedback and guide the operator to exert and maintain the TARGET cricoid pressure during rapid sequence induction (RSI).

In this study we aim to verify the sensor system with a manikin and compare the forces applied by nurses with the sensor system and without.

DETAILED DESCRIPTION:
A total of 22 nurses or anesthetists will be recruited Inclusion criteria include healthy subjects Exclusion criteria include (1) pregnant subjects (2) history of back pain or injury

Cricoid pressure applied on manikin will be measured

1. By electronic medical grade weighing scale
2. By sensor system electronically

ELIGIBILITY:
Inclusion Criteria:

- Healthy status

Exclusion Criteria:

* Pregnant state
* History of problems/ surgery to neck or spine.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05-01; Primary Completion 2016-10-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Force applied (Newton) within targeted range | Each application of cricoid pressure of 60 seconds
  % target cricoid force achieved with and without using cricoid force sensor system
Average force applied during application of 60 seconds | Each application of cricoid pressure of 60 seconds
  Measurement with electronic weighing system and force sensor system

SECONDARY OUTCOMES:
Repeatability of force applied | Minimum 2 weeks apart
  Measurement with electronic weighing system and cricoid force sensor system
Consistency in measurements between cricoid force system and electronic wee | Each application of cricoid pressure of 60 seconds
  Difference in Measurement with electronic weighing system and cricoid force sensor system
User performance over time | Each application of cricoid pressure of 60 seconds
  Cricoid force achieved with time during cricoid force application

OTHER OUTCOMES:
Usability evaluation of cricoid force sensor system | 1 day
  Usability questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- KKWH, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes